CLINICAL TRIAL: NCT02963493
Title: A Single Arm, Open-Label, Phase 2 Study of Melflufen in Combination With Dexamethasone in Patients With Relapsed Refractory Multiple Myeloma Who Are Refractory to Pomalidomide and/or an Anti-CD38 Monoclonal Antibody
Brief Title: A Study of Melphalan Flufenamide (Melflufen) Plus Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Acronym: HORIZON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncopeptides AB (Industry)
Collaborators: Precision For Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OP-106
Record Dates: First submitted 2016-10-18; First posted 2016-11-15 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma
Keywords: relapsed refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — L-melphalanyl-p-L-fluorophenylalanine ethyl ester; melflufen; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- melphalan flufenamide (melflufen) + dexamethasone (Experimental): Melphalan flufenamide (melflufen) 40 mg Day 1 and dexamethasone 40 mg (20 mg for patients 75 years or older) on Days 1, 8, 15 and 22 of each 28-day cycle.
  Interventions: Drug: Melphalan flufenamide (Melflufen); Drug: Dexamethasone

INTERVENTIONS:
Drug: Melphalan flufenamide (Melflufen)
  Other Names: Pepaxto
Drug: Dexamethasone — IV dexamethasone may be substituted for oral dexamethasone in the US. Oral only in Europe.

SUMMARY:
This study will evaluate melflufen in combination with dexamethasone in adult patients with relapsed or refractory multiple myeloma in whose disease is refractory to pomalidomide and/or an anti-CD38 monoclonal antibody. All patients in the study will be treated with melflufen on Day 1 and dexamethasone on Days 1, 8, 15 and 22 of each 28-day cycle.

DETAILED DESCRIPTION:
Melphalan flufenamide (melflufen) is a peptide-drug conjugate that rapidly delivers an alkylating payload into tumor cells. Peptidases are expressed in several cancers, including solid tumors and hematologic malignancies. Melphalan flufenamide is rapidly taken up by myeloma cells due to its high lipophilicity. Once inside the myeloma cell, the activity of melphalan flufenamide is determined by its immediate cleavage by peptidases into hydrophilic alkylator payloads that are entrapped. Melphalan flufenamide is 50-fold more potent than melphalan in myeloma cells in vitro due to increased intracellular alkylator concentration. It rapidly induces irreversible DNA damage leading to apoptosis of myeloma cells. Melphalan flufenamide displays cytotoxic activity against myeloma cell lines resistant to other treatments, including alkylators, in vitro. Melphalan flufenamide also has demonstrated inhibition of angiogenesis and DNA damage with a lack of functional DNA repair in preclinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older
* A prior diagnosis of multiple myeloma with documented disease progression
* Measurable disease based on either of a) serum monoclonal protein by protein electrophoresis (SPEP), b) monoclonal protein in the urine on 24-hour urine electrophoresis (UPEP), and/or c) serum immunoglobulin free light chain combined with abnormal serum immunoglobulin kappa to lambda free light chain ratio
* A minimum of 2 prior lines of therapy including an IMiD and a PI and is refractory to pomalidomide and/or daratumumab
* Life expectancy of ≥ 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Female of child bearing potential (FCBP) and non-vasectomized male agree to practice appropriate methods of birth control
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information
* 12-lead ECG with QTc interval within defined limit
* Acceptable laboratory results during screening and prior to first study drug administration of the following parameters: absolute neutrophil count (ANC), platelet count, hemoglobin, total bilirubin, aspartate transaminase (AST/SGOT) and alanine transaminase (ALT/SGPT), renal function based on estimated creatinine clearance
* Must have, or accept to have, an acceptable central catheter for infusion of melflufen

Exclusion Criteria:

* Evidence of mucosal or internal bleeding and/or is platelet transfusion refractory
* Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient or would adversely affect his/her participating in this study
* Known active infection requiring parenteral or oral anti-infective treatment within defined period
* Primary refractory disease
* Other malignancy diagnosed or requiring treatment within the defined period with specific exceptions
* Pregnant or breast-feeding females
* Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse compliance or follow-up evaluation
* Known HIV or active hepatitis B or C viral infection
* Concurrent symptomatic amyloidosis or plasma cell leukemia
* POEMS syndrome [plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes]
* Previous cytotoxic therapies, including cytotoxic investigational agents, for multiple myeloma within defined values prior to start of study treatment
* Residual side effects to previous therapy over specific grade prior to initiation of therapy
* Prior autologous or allogeneic stem cell transplant within defined period of initiation of therapy
* Prior allogeneic stem cell transplant with active graft-versus-host- disease (GVHD).
* Prior major surgical procedure or radiation therapy within specified period of the first dose of study treatment (with defined exception).
* Known intolerance to steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Harmenberg, MD, PhD, Study Chair — Oncopeptides AB
Locations (20):
- United States (9):
  - Innovative Clinical Research Institute (ICRI), Whittier, California
  - University of Florida, Gainesville, Florida
  - RUSH, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Hudson Valley Hematology Oncology, Poughkeepsie, New York
  - UPMC Hillman Cancer Insitute, Pittsburgh, Pennsylvania
  - Baylor, Dallas, Texas
- France (2):
  - CHU de Nantes, Nantes
  - CHU de Poitiers, Poitiers
- Italy (2):
  - Universita di Bolognia, Bologna
  - Turin Hospital Myeloma Unit, Turin
- Spain (7):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Institut Català d'Oncología (ICO) Badalona, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Complejo Hospitalario de Salamanca, Salamanca
  - Hospital Universitario Doctor Peset, Valencia

REFERENCES:
- [Result] Richardson PG, Oriol A, Larocca A, Blade J, Cavo M, Rodriguez-Otero P, Leleu X, Nadeem O, Hiemenz JW, Hassoun H, Touzeau C, Alegre A, Paner A, Maisel C, Mazumder A, Raptis A, Moreb JS, Anderson KC, Laubach JP, Thuresson S, Thuresson M, Byrne C, Harmenberg J, Bakker NA, Mateos MV; HORIZON (OP-106) Investigators. Melflufen and Dexamethasone in Heavily Pretreated Relapsed and Refractory Multiple Myeloma. J Clin Oncol. 2021 Mar 1;39(7):757-767. doi: 10.1200/JCO.20.02259. Epub 2020 Dec 9. PMID 33296242
- [Derived] Sonneveld P, Richardson PG, Ludwig H, Dimopoulos MA, Schjesvold FH, Hajek R, Abdulhaq H, Thuresson M, Norin S, Bakker NA, Mateos MV. Benefit Versus Risk Assessment of Melflufen and Dexamethasone in Relapsed/Refractory Multiple Myeloma: Analyses From Longer Follow-up of the OCEAN and HORIZON Studies. Clin Lymphoma Myeloma Leuk. 2023 Sep;23(9):687-696. doi: 10.1016/j.clml.2023.05.004. Epub 2023 May 6. PMID 37355418
- [Derived] Larocca A, Leleu X, Touzeau C, Blade J, Paner A, Mateos MV, Cavo M, Maisel C, Alegre A, Oriol A, Raptis A, Rodriguez-Otero P, Mazumder A, Laubach J, Nadeem O, Sandberg A, Orre M, Torrang A, Bakker NA, Richardson PG. Patient-reported outcomes in relapsed/refractory multiple myeloma treated with melflufen plus dexamethasone: analyses from the Phase II HORIZON study. Br J Haematol. 2022 Feb;196(3):639-648. doi: 10.1111/bjh.17887. Epub 2021 Oct 21. PMID 34671975

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 157 Patients were enrolled and treated on study
Groups:
- Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set: Melphalan flufenamide (melflufen) 40 mg Day 1 and dexamethasone 40 mg (reduced dose for patients 75 years or older) on Days 1, 8, 15 and 22 of each 28-day cycle.
  Melphalan flufenamide (Melflufen)
  Dexamethasone
Period: Overall Study
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set
Started | 157
Completed (Study completion for assessment of endpoints) | 157
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Melphalan Flufenamide (Melflufen) + Dexamethasone: Melphalan flufenamide (melflufen) 40 mg Day 1 and dexamethasone 40 mg (reduced dose for patients 75 years or older) on Days 1, 8, 15 and 22 of each 28-day cycle.
  Melphalan flufenamide (Melflufen)
  Dexamethasone
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone
Number analyzed (Participants) | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 78
  >=65 years | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 137
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 11
  White | 132
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 69
  Italy | 23
  France | 13
  Spain | 52
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status Categories Status 0: Normal activity, fully active, able to carry on all pre-disease performance without restriction.
  Status 1: Symptoms, but fully ambulatory, restricted in physically strenuous but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Status 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Status 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours.
  Participants
    Performance Status 0 | 39
    Performance Status 1 | 93
    Performance Status 2 | 24
    Performance Status 3 | 1
Weight [Mean (Standard Deviation); unit: kilograms] — Population: Baseline weight not recorded for one patient
  kilograms
    number analyzed (Participants) | 156
    (all) | 74.3 (17.41)
International Staging System (ISS) [Count of Participants; unit: Participants] — International Staging System (ISS) is an assessment of risk factors for multiple myeloma ISS Stage I: Serum B2-microglobulin < 3.5 mg/L, serum albumin ≥ 3.5 g/dL ISS Stage II: Not ISS Stage I or III ISS Stage III: Serum B 2-microglobulin ≥ 5.5 mg/L
  Participants
    International Staging System (ISS) Stage I | 63
    International Staging System (ISS) Stage II | 49
    International Staging System (ISS) Stage III | 39
    Unknown | 4
    Missing | 2
Time since initial diagnosis [Mean (Standard Deviation); unit: years] | 7.0 (3.46)
Extramedullary disease at study entry [Count of Participants; unit: Participants] | 55
Type of measurable disease at baseline [Count of Participants; unit: Participants] — Serum M-protein ≥ 0.5 g/dL (SPEP), urine M-protein ≥ 200 mg/24 hours (UPEP), or serum free light chain (sFLC) assay with FLC ≥ 10 mg/dL (≥ 100 mg/L) and abnormal serum immunoglobulin kappa to lambda FLC ratio. Population: 5 patients did not have all assessments completed to adequately categorize
  Participants
    SPEP and UPEP | 33
    SPEP only | 63
    UPEP only | 37
    sFLC only | 20
    Unable to determine | 4
Cytogenetic risk group based on FISH at study entry [Count of Participants; unit: Participants] — High-risk cytogenetic abnormalities at study entry is defined as patients who had the genetic subtype t(4; 14), t(14:16), deletion 17p, gain 1q (+1q), or t(14,20) determined by Baseline fluorescence in situ hybridization (FISH)
  Participants
    High | 59
    Standard | 67
    Unknown | 31
Heavy-light chain combination at study entry [Count of Participants; unit: Participants]
  IgA-Kappa | 18
  IgA-Lambda | 12
  IgD-Kappa | 1
  IgD-Lambda | 1
  IgG-Kappa | 57
  IgG-Lambda | 31
  IgM-Kappa | 2
  Multiple-Kappa | 2
  None-Kappa | 19
  None-Lambda | 13
  Unknown-Kappa | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The overall response rate (ORR) will be estimated as the percentage of patients who achieve sCR, CR, VGPR, or PR as their best response as assessed by the investigator. Response assessed by IMWG (International myeloma working group) criteria sCR-stringent complete response: CR plus Normal FLC (free light chain) ratio and absence of clonal cells in BM CR-complete response: Negative immunofixation in serum/urine; Disappearance of soft tissue plasmacytomas; <5% plasma cells in BM; If only FLC disease, normal FLC ratio (0.26-1.65) VGPR-very good partial response: Serum/urine M-protein detectable by immunofixation but not electrophoresis or ≥90% reduction in serum M-protein and urine M-protein <100 mg/24 h; If only FLC disease, >90% decrease in the difference between involved and uninvolved FLC levels PR-partial response: 50% reduction of serum M-protein and soft tissue plasmacytomas, ≥90% reduction in urinary M-protein or to <200 mg/24 h; other special cases if M-protein unmeasurable
Time Frame: Patients were followed until documented progression, unacceptable toxicity, patient/physician decision to withdraw or date of death, whichever came first. Longest time to response in study recorded as 15.3 months. Longest time on treatment 35 months.
Measure: Count of Participants; unit: Participants
Groups:
- Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set: Full analysis set
  Melphalan flufenamide (melflufen) 40 mg Day 1 and dexamethasone 40 mg (reduced dose for patients 75 years or older) on Days 1, 8, 15 and 22 of each 28-day cycle.
  Melphalan flufenamide (Melflufen)
  Dexamethasone: IV dexamethasone may be substituted for oral dexamethasone in the US. Oral only in Europe.
- Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Extramedullary Disease: Patients with extramedullary disease at baseline defined as myeloma disease either originating in, but extending beyond, the cortical bone or as a separate soft tissue mass
- Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease: Triple class refractory population defined as refractory to or intolerant of at least one immunomodulatory drug, at least one proteasome inhibitor, and at least one anti-CD38 monoclonal antibody
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Extramedullary Disease | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease
Number analyzed (Participants) | 157 | 55 | 119
Participants | 53 | 14 | 35

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from start of treatment to either progression or death, whichever comes first as assessed by the investigator using IMWG criteria. Progression of disease is defined by an increase of 25% from the lowest response for either of Serum M-component (absolute increase of ≥ 0.5 g/dL) or Urine M-component (absolute increase of ≥200 mg/ 24h); In patients without measurable M-protein a 25% increase in the difference between involved and uninvolved FLC (free light chain) levels (absolute increase must be >10 mg/dL); If unmeasurable FLC levels, a 25% increase in bone marrow plasma cell percentage (absolute percentage must be >10%); New bone or soft tissue plasmacytomas or definite increase in existing ones; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the plasma cell proliferative disorder
Time Frame: Patients were followed until documented progression, unacceptable toxicity, patient/physician decision to withdraw or date of death, whichever came first. Longest follow-up time for PFS recorded as 37.2 months at study end.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set: Melphalan flufenamide (melflufen) 40 mg Day 1 and dexamethasone 40 mg (reduced dose for patients 75 years or older) on Days 1, 8, 15 and 22 of each 28-day cycle.
  Melphalan flufenamide (Melflufen)
  Dexamethasone: IV dexamethasone may be substituted for oral dexamethasone in the US. Oral only in Europe.
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Extramedullary Disease | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease
Number analyzed (Participants) | 157 | 55 | 119
months | 4.27 [3.42 to 4.90] | 2.89 [1.97 to 3.94] | 3.94 [3.09 to 4.67]

3. Secondary Outcome: Duration of Response
Description: Time from first response to progression based on investigator assessment. See definitions of response and progression in ORR and PFS outcomes.
Time Frame: From date of response until the date of first documented progression or date of death from any cause, whichever came first. Longest time of response recorded as 36.2 months at study end.
Population: Patients with a best response of PR or better as determined by the investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Extramedullary Disease | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease
Number analyzed (Participants) | 47 | 15 | 31
months | 6.90 [4.40 to 10.38] | 5.49 [2.10 to 12.71] | 7.46 [4.24 to 10.38]

4. Secondary Outcome: Overall Survival
Description: Time from start of treatment to death
Time Frame: From date of first dose of study medication until the date of death from any cause, assessed up to 24 months after study drug discontinuation.
Population: Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Extramedullary Disease | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease
Number analyzed (Participants) | 157 | 55 | 119
months | 11.79 [9.53 to 14.55] | 6.44 [5.06 to 9.66] | 10.12 [7.20 to 12.29]

5. Secondary Outcome: Functional Status and Well-being: EORTC QLQ-C30
Description: Change from baseline in Patient Reported Outcome questionnaire EORTC QLQ-C30. The EORTC QLQ-C30 includes 30 items resulting in 5 functional scales, 1 Global Health Status scale, 3 symptom scales, and 6 single items. The recall period is 1 week (the past week). The scales are transformed to a 0 (worst) to 100 (best) scale. The QLQ-C30 summary score is calculated as the mean of the combined 13 QLQ-C30 scale and item scores (excluding global QoL and financial impact), with a higher score indicating a better HRQoL. If at least 50% of the items from the scale had been answered, the missing items were assumed to have values equal to the average of those items which were present for that respondent.
Time Frame: To be assessed prior to dosing at Cycle 1, 2, 4, 6, 8, and End of Treatment. 23 patients were ongoing for QoL assessments at data cutoff. QoL was added in Protocol Amendment 4 beginning in Oct. 2018.
Population: This outcome measure was prespecified to be analyzed/reported for the Mel + Dex: FAS Arm/Group and Mel + Dex: Patients With TCR Disease.
  62 pts in the FAS included after QoL was added in Amd 4, whereof 48 pts in the sub-group of pts with TCR disease.
  This outcome measure was not analyzed/reported separately for the sub-group of patients with EMD as there were limited no. of pts with EMD among the QoL patients. No data/results are available to report for patients with EMD.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease
Number analyzed (Participants) | 62 | 48
units on a scale
  Baseline value | 75.5 (13.2) | 74.9 (13.0)
  Cycle 2 Day 1 Change from baseline: number analyzed (Participants) | 51 | 39
  Cycle 2 Day 1 Change from baseline | 0.2 (11.9) | 74.8 (13.7)
  Cycle 4 Day 1 Change from baseline: number analyzed (Participants) | 36 | 27
  Cycle 4 Day 1 Change from baseline | -2.6 (12.8) | 76.9 (11.9)
  Cycle 6 Day 1 Change from baseline: number analyzed (Participants) | 21 | 14
  Cycle 6 Day 1 Change from baseline | -3.3 (11.5) | 73.2 (12.6)
  Cycle 8 Day 1 Change from baseline: number analyzed (Participants) | 13 | 9
  Cycle 8 Day 1 Change from baseline | -7.5 (10.6) | 71.3 (11.3)

6. Secondary Outcome: Functional Status and Well-being: EQ-5D-3L
Description: Change from baseline in Patient Reported Outcome questionnaire EQ-5D-3L. The EQ-5D-3L questionnaire converts 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression of patient-reported, current-day health status into a "health utility" score. For the EQ-5D-3L questionnaire, each dimension is scored on an ordinal scale with 3 available levels of response and scores ranging from 1 to 3, "no problems," "some problems," and "extreme problems," respectively. The EQ VAS scores rates "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). No imputation of missing items or composite scores were done. The scores for the 5 dimensions are used to compute a single utility score ranging from zero (0.0) to 1 (1.0) representing the general health status of the individual.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Change in composite scale score
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease
Number analyzed (Participants) | 62 | 48
Change in composite scale score
  Baseline value | 0.6748 (0.2243) | 0.6803 (0.2086)
  Cycle 2 Day 1 Change from baseline: number analyzed (Participants) | 62 | 37
  Cycle 2 Day 1 Change from baseline | -0.0228 (0.1848) | -0.0502 (0.1846)
  Cycle 4 Day 1 Change from baseline: number analyzed (Participants) | 34 | 25
  Cycle 4 Day 1 Change from baseline | -0.0169 (0.2187) | 0.0038 (0.1919)
  Cycle 6 Day 1 Change from baseline: number analyzed (Participants) | 18 | 11
  Cycle 6 Day 1 Change from baseline | -0.0786 (0.3049) | -0.1486 (0.3309)
  Cycle 8 Day 1 Change from baseline: number analyzed (Participants) | 14 | 9
  Cycle 8 Day 1 Change from baseline | -0.1461 (0.2320) | -0.2174 (0.2464)
  End of Treatment Change from baseline: number analyzed (Participants) | 31 | 26
  End of Treatment Change from baseline | -0.0014 (0.2594) | 0.0124 (0.2552)

7. Secondary Outcome: Clinical Benefit Rate
Description: The clinical benefit rate (CBR) will be estimated as the percentage of patients who achieve sCR, CR, VGPR, PR, or MR as their best response as assessed by the investigator. See Primary Outcome (ORR) for definitions of response categories.
Time Frame: Patients were followed until documented progression, unacceptable toxicity, patient/physician decision to withdraw or date of death, whichever came first. Longest time on study treatment recorded as 35.0 months at study end.
Measure: Count of Participants; unit: Participants
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Extramedullary Disease | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease
Number analyzed (Participants) | 157 | 55 | 119
Participants | 72 | 17 | 48

8. Secondary Outcome: Time to Response
Description: Duration from start of treatment to the first occurrence of a confirmed response of PR or better as assessed by the investigator. See definitions of response in Primary Outcome (ORR).
Time Frame: From start of treatment to first confirmed response. Longest time to response in study recorded as 15.3 months.
Population: This outcome measure was pre-specified to be analyzed/reported for the Mel + Dex: FAS Arm/Group and "Mel + Dex: Patients With TCR Disease.
  This outcome measure was analyzed/reported for patients with a best response of PR or better in the full analysis set as well as in the sub-group of patients with triple class refractory disease.
  This outcome measure was not analyzed/reported separately for the sub-group of patients with Extramedullary Disease. No data available to report for EMD patients.
Measure: Median (Full Range); unit: months
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease
Number analyzed (Participants) | 53 | 35
months | 2.1 [1.0 to 15.3] | 2.1 [1.0 to 15.3]

9. Secondary Outcome: Time to Progression
Description: Duration from start of treatment to first evidence of disease progression as assessed by the investigator. See definitions of response and progression in ORR and PFS outcomes.
Time Frame: From start of treatment to first evidence of disease progression or date of death from any cause, whichever came first. Longest time to progression recorded was 37.2 months at study end.
Population: This outcome measure was prespecified to be analyzed/reported for the Mel + Dex: FAS Arm/Group and Mel + Dex: Patients With TCR Disease.
  This outcome measure was analyzed/reported for patients in the full analysis set as well as in the sub-group of patients with triple class refractory disease.
  This outcome measure was not analyzed/reported separately for the sub-group of patients with Extramedullary Disease. No data available to report for EMD patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease
Number analyzed (Participants) | 157 | 119
months | 4.4 [3.71 to 5.32] | 4.11 [3.32 to 4.86]

ADVERSE EVENTS:
Time Frame: Patients were treated in 28 day cycles indefinitely until withdrawal from study, with the longest time on study of 17 months. Adverse events were collected until 30 days after the last dose of study drug. Patients were followed for survival for 24 months after disease progression or start of subsequent anti-myeloma therapy.
Description: The Safety Analysis Set for evaluation of adverse events included all patients who received at least one dose of melflufen or dexamethasone in the study. Patients that were triple-class refractory and those with extramedullary disease were defined as a subgroups of interest for evaluation.
Arm/Group | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Extramedullary Disease | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease
All-Cause Mortality (participants affected / at risk) | 130/157 | 51/55 | 105/119
Serious Adverse Events (participants affected / at risk) | 88/157 | 38/55 | 70/119
Other Adverse Events (participants affected / at risk) | 157/157 | 55/55 | 119/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set (N=157) | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Extramedullary Disease (N=55) | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease (N=119)
Pneumonia (Infections and infestations) | 16 (16) | 6 (6) | 8 (8)
Respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 4 (4)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (10) | 3 (4) | 6 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 3 (4) | 5 (6)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 5 (5) | 4 (4) | 5 (5)
Pyrexia (General disorders) | 3 (4) | 1 (2) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 2 (3) | 4 (5)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 4 (6) | 2 (2) | 4 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (5) | 3 (4) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (3) | 2 (3) | 2 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fungal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Lower respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 3 (4) | 3 (4) | 3 (4)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (2) | 1 (2) | 1 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 | 0
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Face oedema (General disorders) | 1 (1) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiac amyloidosis (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperammonaemic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 1 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 3 (3)
Refractory cytopenia with multilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerecrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan Flufenamide (Melflufen) + Dexamethasone: Full Analysis Set (N=157) | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Extramedullary Disease (N=55) | Melphalan Flufenamide (Melflufen) + Dexamethasone: Patients With Triple Class Refractory Disease (N=119)
Anaemia (Blood and lymphatic system disorders) | 113 (432) | 35 (154) | 78 (300)
Thrombocytopenia (Blood and lymphatic system disorders) | 93 (628) | 27 (130) | 64 (415)
Neutropenia (Blood and lymphatic system disorders) | 86 (549) | 23 (126) | 60 (374)
Leukopenia (Blood and lymphatic system disorders) | 12 (53) | 3 (11) | 9 (41)
Lymphopenia (Blood and lymphatic system disorders) | 8 (77) | 3 (44) | 6 (65)
Fatigue (General disorders) | 46 (74) | 14 (24) | 35 (56)
Asthenia (General disorders) | 45 (73) | 11 (22) | 30 (50)
Pyrexia (General disorders) | 39 (64) | 9 (11) | 28 (49)
Oedema peripheral (General disorders) | 23 (25) | 9 (11) | 12 (14)
Nausea (Gastrointestinal disorders) | 51 (67) | 16 (19) | 39 (53)
Diarrhoea (Gastrointestinal disorders) | 43 (67) | 14 (21) | 28 (45)
Constipation (Gastrointestinal disorders) | 24 (26) | 11 (13) | 20 (22)
Vomiting (Gastrointestinal disorders) | 23 (30) | 10 (12) | 20 (26)
Abdominal pain (Gastrointestinal disorders) | 10 (15) | 6 (11) | 6 (11)
Upper respiratory tract infection (Infections and infestations) | 24 (43) | 13 (25) | 19 (35)
Pneumonia (Infections and infestations) | 6 (7) | 3 (3) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 21 (24) | 8 (10) | 15 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 (26) | 12 (12) | 18 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (21) | 6 (7) | 11 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (25) | 7 (12) | 13 (15)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 4 (7) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 7 (9) | 9 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 4 (5) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (38) | 8 (9) | 21 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 7 (8) | 16 (20)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 7 (7) | 11 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (19) | 6 (10) | 12 (17)
Decreased appetite (Metabolism and nutrition disorders) | 22 (25) | 6 (7) | 13 (16)
Hypokalaemia (Metabolism and nutrition disorders) | 23 (39) | 9 (15) | 16 (25)
Hypocalcaemia (Metabolism and nutrition disorders) | 17 (27) | 6 (10) | 11 (18)
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 (28) | 7 (14) | 11 (18)
Hypophosphataemia (Metabolism and nutrition disorders) | 14 (25) | 6 (11) | 10 (18)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (15) | 2 (2) | 7 (7)
White blood cell count decreased (Investigations) | 45 (175) | 20 (78) | 35 (138)
Neutrophil count decreased (Investigations) | 42 (210) | 20 (83) | 33 (166)
Platelet count decreased (Investigations) | 40 (151) | 19 (56) | 33 (129)
Blood creatinine increased (Investigations) | 10 (17) | 1 (2) | 7 (13)
Headache (Nervous system disorders) | 21 (22) | 6 (7) | 17 (18)
Dizziness (Nervous system disorders) | 18 (22) | 1 (1) | 9 (13)
Insomnia (Psychiatric disorders) | 18 (22) | 4 (5) | 12 (13)
Hypotension (Vascular disorders) | 8 (12) | 3 (6) | 6 (10)
Contusion (Injury, poisoning and procedural complications) | 17 (25) | 7 (9) | 13 (19)
Tachycardia (Cardiac disorders) | 9 (12) | 6 (9) | 8 (11)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 3 (4) | 6 (7)
Weight decreased (Investigations) | 7 (7) | 5 (5) | 7 (13)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (9) | 2 (2) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 1 (1) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT02963493/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT02963493/SAP_002.pdf